CLINICAL TRIAL: NCT06590792
Title: Relationship Between Oxidative Stress and Aortic Stiffness During Acute Exhaustive Training in Adolescent Football Players
Brief Title: Relationship Between Oxidative Stress and Aortic Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Şensu Dinçer, medical doctor, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Soccer aortic stiffness
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Aortic Stiffness; Oxidative Stress; Football Player
Keywords: stiffness; elastography; football; oxidative stress

STUDY DESIGN:
Intervention Model Description: Two groups including 20 participants in each of them will be involved the study. One group will consist of adolescent football players, while the other group will consist of non-athlete healthy participants
Who Masked: Investigator, Outcomes Assessor
Masking Description: Echocardiographer and biochemistry expert will be blind to participants type (sedentary or football player)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- football player (Experimental): 14-18 years old male football players who play in the infrastructure of a football club
  Interventions: Other: exhaustive exercise training session
- healthy control group (Active Comparator): 14-18 years old male healthy participants who don't involve any regular sports training
  Interventions: Other: exhaustive exercise training session

INTERVENTIONS:
Other: exhaustive exercise training session — Cardiovascular exercise test will be performed by the participants. This test is sustained until the participants feel exhausted.

SUMMARY:
The goal of this clinical trial is to search about if there is any relationship between the aortic stiffness and oxidative stress response in adolescent football players. The main questions are;

* Is there any difference between the adolescent football players and healthy sedentary control group in terms of oxidative stress and aortic stiffness parameters?
* Is there any relationship between the aortic stiffness and oxidative response to acute exercise training in adolescent male football players? Participants will perform acute exhaustive exercise training. Venous blood will be drained before and after exercise training. Oxidative parameters will be measured.

DETAILED DESCRIPTION:
Arterial stiffness is defined as stiffening of the arterial wall and refers to a decrease in the capacity of an artery to expand and contract in response to pressure changes in the vessel. The parameters indicating arterial stiffness are compliance and distensibility of the vessel.

Imbalance in the formation of vasodilator and vasoconstrictor signaling molecules acting on the vessel is an important determining factor in the development of endothelial dysfunction, which is often exacerbated by oxidative stress. Disruption of the balance between oxidants and antioxidants in favor of oxidants leads to disruption of the elastin-collagen ratio in the vessel wall in favor of collagen and ultimately to the development of arterial stiffness. Regular exercise is beneficial both to prevent the development of arterial stiffness and to reduce arterial stiffness. Although many mechanisms have been mentioned for exercise to improve endothelial function, there is no clear consensus on the mechanisms by which exercise increases arterial compliance, which is one of the indicators of atherosclerosis. While the beneficial impacts of physical activity on arterial stiffness are well-documented, this varies considerably among sports disciplines. For instance, there are studies showing that endurance training decreases arterial stiffness in young adults and elderly individuals, whereas strength training increases arterial stiffness. Arterial stiffness is lower in endurance athletes with a longer sports history and higher in those with a strength training history. The weekly training time of competitive young athletes is well beyond the amount of exercise required for healthy living. It has also been suggested that this excessive amount of time may trigger some unfavorable adaptations in the cardiovascular system. In addition, the number of studies examining the effects of regular exercise training at these levels on the vascular system is limited. Studies indicate that changes in arterial stiffness start at early ages and this is also true for young athletes who perform regular training in the infrastructures of various sports branches. Therefore, our aim is investigating the relationship between the oxidative stress parameters and aortic stiffness in adolescent male football players and comparing with the healthy control group. Secondly, the investigators will evaluate if there is any difference between the aortic stiffness and oxidative response to acute exercise training in adolescent male football players?

ELIGIBILITY:
Inclusion Criteria:

* age between 14-18
* male gender
* football player
* attending regular football training for at least 1 season

Exclusion Criteria:

* female gender
* attending any other sports training except from football
* having any chronic disease
* having any musculoskeletal disease which limits to join exhaustive exercise training

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
aortic strain (%) | will be measured twice before and after acute exhaustive exercise, through study completion, up to 8 weeks
  =[(aortic systolic diameter - diastolic diameter)× 100] / aortic diastolic diameter
aortic stiffness index | will be measured twice before and after acute exhaustive exercise,through study completion, up to 8 weeks
  = ln (systolic pressure / diastolic pressure) / aortic strain
aortic distensibility (cm2.dyn-1.10-6) | will be measured twice before and after acute exhaustive exercise,through study completion, up to 8 weeks
  = (2 × aortic strain) / (systolic pressure-diastolic pressure)
serum lipid hydroperoxide assay | will be measured twice before and after acute exhaustive exercise,through study completion, up to 8 weeks
  lipid hydroperoxide (LHP) level of serum (nmol/mL). Lipid hydroperoxide (LOOH) is the first, comparatively stable, product of the lipid peroxidation reaction.
serum malondialdehide assay | will be measured twice before and after acute exhaustive exercise,through study completion, up to 8 weeks
  serum malondialdehide (MDA) level of serum (nmol/mL).MDA is the end product of the oxidation of polyunsaturated fatty acids.
serum advanced oxidation protein products assay | will be measured twice before and after acute exhaustive exercise,through study completion, up to 8 weeks
  Advanced oxidation protein products (AOPP) level of serum (mikromol/L ). AOPP are the dityrosine-containing and crosslinking protein products formed during oxidative stress by reaction of plasma protein with chlorinated oxidants, and often carried by albumin in vivo
serum advanced glycation end products assay | will be measured twice before and after acute exhaustive exercise,through study completion, up to 8 weeks
  serum advanced glycation end products (AGE) level of serum(FU/mg). AGEs are are a heterogeneous group of proteins and lipids, formed by nonenzymatic glycation after persistent contact with aldose sugars
serum ferric reducing antioxidant power assay | will be measured twice before and after acute exhaustive exercise, through study completion, up to 8 weeks
  ferric reducing antioxidant power (FRAP) level of serum (mikromol/mL ). FRAP is an antioxidant capacity assay that uses Trolox as a standard
serum superoxide dismutase activity assay | will be measured twice before and after acute exhaustive exercise,through study completion, up to 8 weeks
  copper-zinc superoxide dismutase activity (SOD) level of serum (U/mL). SODs are enzymes that catalyze the conversion of naturally-occuring but harmful superoxide radicals into molecular oxygen and hydrogen peroxide
serum total antioxidant status and total oxidant status assay | will be measured twice before and after acute exhaustive exercise,through study completion, up to 8 weeks
  total antioxidant status (TAS) and total oxidant status (TOS) levels of serum (trolox equivalent/L) are two indicators to determine all antioxidants or oxidants in samples, which can more comprehensively reflect the changes of oxidant and antioxidant capacity of samples

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Faculty of Medicine, Istanbul
  - Şensu Dinçer, Istanbul